CLINICAL TRIAL: NCT06676319
Title: A Randomized, Phase 2, Double-blind, Placebo-controlled, Parallel-group, 2-arm Study to Investigate the Efficacy, Safety, and Tolerability of Subcutaneous Lunsekimig (SAR443765) in Adult Participants With High-risk Asthma Who Are Not Currently Eligible for Biologic Treatment
Brief Title: Study of Lunsekimig (SAR443765) Compared With Placebo in Adults With High-risk Asthma
Acronym: AIRLYMPUS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ACT18301; 2024-513959-33 (Registry Identifier: CTIS); U1111-1301-3938 (Registry Identifier: ICTRP)
Record Dates: First submitted 2024-11-04; First posted 2024-11-06 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Fluticasone-Salmeterol Drug Combination; Budesonide, Formoterol Fumarate Drug Combination; Budesonide; Albuterol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Lunsekimig (Experimental): Participants will receive lunsekimig (SC injection) every 4 weeks
  Interventions: Drug: Lunsekimig; Drug: Short-Acting Beta Agonists (SABA); Drug: Fluticasone/Salmeterol; Drug: Budesonide/Formoterol; Drug: Budesonide/Albuterol
- Placebo (Placebo Comparator): Participants will receive placebo (SC injection) every 4 weeks
  Interventions: Drug: Short-Acting Beta Agonists (SABA); Drug: Placebo; Drug: Fluticasone/Salmeterol; Drug: Budesonide/Formoterol; Drug: Budesonide/Albuterol

INTERVENTIONS:
Drug: Lunsekimig — Pharmaceutical form: Solution for injection in vial; Route of administration: Subcutaneous injection
  Other Names: SAR443765
  Arms: Lunsekimig
Drug: Short-Acting Beta Agonists (SABA) — Pharmaceutical form: Varies and depends on pharmaceutical presentation; Route of administration: Oral Inhalation
Drug: Placebo — Pharmaceutical form: Solution for injection in vial; Route of administration: Subcutaneous injection
  Arms: Placebo
Drug: Fluticasone/Salmeterol — Pharmaceutical form: Varies and depends on pharmaceutical presentation; Route of administration:Oral Inhalation
Drug: Budesonide/Formoterol — Pharmaceutical form: Varies and depends on pharmaceutical presentation; Route of administration: Oral Inhalation
Drug: Budesonide/Albuterol — Pharmaceutical form: Aerosol for inhalation; Route of administration: Oral Inhalation

SUMMARY:
This is a parallel-group, Phase 2, randomized, double-blind, placebo-controlled, 2-arm study for the treatment of asthma.

The purpose of this study is to assess the efficacy, safety, and tolerability of add-on therapy with subcutaneous (SC) lunsekimig compared with placebo in male and female participants (aged 18 to 80 years, inclusive) with asthma, who are not currently eligible for biologic treatments.

Study details include:

* The study duration will be approximately 64 weeks for participants not transitioning into the LTS study and approximately 60 weeks for participants transitioning into the LTS study.
* The investigational treatment duration will be up to approximately 52 weeks.
* The number of visits will be 18.

ELIGIBILITY:
Inclusion Criteria:

* Physician-diagnosed mild-to-moderate asthma for more than 12 months based on GINA guidelines.
* At least 1 asthma exacerbation in the year prior to Screening (Visit 1).
* Pre-BD FEV1 of equal or more than 40% of predicted normal (by Global Lung Function Initiative [GLI] standards) at Screening (Visit 1).

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

* Other severe lung diseases (eg, chronic obstructive pulmonary disease [COPD]. bronchiectasis, idiopathic pulmonary fibrosis, etc) which may impair lung function.
* Participants who experience a deterioration of asthma that results in emergency treatment or hospitalization, or treatment with systemic steroids within 1 month prior to the Screening (Visit 1) (counting from the date of completion of treatment for asthma exacerbation).
* Participants who have experienced an upper or lower respiratory tract infection within the 4 weeks prior to Screening (Visit 1).
* Known history of, or suspected, significant current immunosuppression, including history of invasive opportunistic or helminthic infections despite infection resolution or otherwise recurrent infections of abnormal frequency or prolonged duration.
* Evidence of any infection requiring systemic anti-infective treatment within 2 weeks before Screening (Visit 1) or during the screening period. Significant viral infections within 2 weeks before Screening (Visit 1) or during the screening period even if the participant has not received systemic antiviral treatment (eg, influenza receiving only symptomatic treatment).
* Participants with active tuberculosis (TB), latent TB, a history of incompletely treated TB, suspected extrapulmonary TB infection, or who are at high risk of contracting TB (such as close contact with individuals with active TB), or received Bacillus Calmette-Guérin (BCG)-vaccination within 12 weeks prior to Screening (Visit 1).
* Severe concomitant illness that would in the Investigator's opinion inhibit the participant's participation in the study, including for example, but not limited to, hypertension, renal disease, neurological conditions, heart failure, and pulmonary disease.

NOTE: The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1147 (Estimated)
Dates: Start 2024-11-07 (Actual); Primary Completion 2027-09-17 (Estimated); Study Completion 2027-10-15 (Estimated)

PRIMARY OUTCOMES:
Annualized rate of asthma exacerbation events | From baseline up to 52 weeks
  Asthma exacerbation event defined as: worsening of asthma requiring the use of systemic corticosteroids for ≥3 days; or hospitalization or emergency room visit due to asthma and requiring the use of systemic corticosteroids or death due to asthma

SECONDARY OUTCOMES:
Change from baseline in prebronchodilator (BD) forced expiratory volume in 1 second (FEV1) | From baseline to week 52
Change from baseline in Asthma Control Questionnaire5 (ACQ-5) score | From baseline to week 52
  The ACQ-5 is a questionnaire that measures the adequacy of asthma control and any changes in asthma control that may occur spontaneously or as a result of treatment. The ACQ-5 has five questions on the asthma symptoms and patients are asked to recall how their asthma has been during the previous week and to respond on a 7-point scale for each question (0 = no impairment, 6 = maximum impairment). The ACQ-5 score is the mean of the 5 questions and, therefore, between 0 (totally controlled) and 6 (severely uncontrolled). A high score indicates low asthma control.
Change from baseline in FeNO level | From baseline to week 52
Annualized rate of loss of asthma control events (LOAC) events | From baseline to week 52
  Annualized rate of LOAC events defined by 1 or more of the following criteria:
  * ≥30% reduction from baseline in morning PEF on 2 consecutive days
  * ≥6 additional reliever puffs of SABA in a 24-hour period (compared to baseline) on 2 consecutive days OR ≥4 additional puffs of low-dose budesonide/formoterol or budesonide/albuterol in a 24-hour period (compared to baseline) on 2 consecutive days
  * Worsening of asthma requiring the use of systemic corticosteroids for ≥3 days
  * Hospitalization or emergency room visit because of asthma, requiring systemic corticosteroids (asthma exacerbation event)
  * Death due to asthma
Annualized rate of asthma exacerbations requiring hospitalization or emergency room or urgent care visit | From baseline to week 52
Total systemic corticosteroid dose exposure | From baseline to week 52
Change from baseline in Asthma Quality of Life Questionnaire Standardized (AQLQ{S}) scores | From baseline to week 52
Change from baseline in the Asthma Daytime Symptom Diary (ADSD) daily morning and evening score | From baseline to week 52
Serum lunsekimig concentrations | From baseline to week 56
Incidence and titer of anti-drug antibodies (ADA) against lunsekimig | From baseline to week 56
Incidence of participants with treatment-emergent adverse events (TEAEs), including local reactions, adverse events of special interests (AESIs), serious adverse events (SAEs) | From baseline to week 56

CONTACTS AND LOCATIONS:
Locations (240):
- United States (58):
  - The Center for Clinical Trials - Saraland- Site Number : 8400096, Saraland, Alabama
  - Chandler Clinical Research Trials- Site Number : 8400075, Chandler, Arizona
  - Epic Medical Research - Sun City- Site Number : 8400052, Sun City, Arizona
  - Tucson Clinical Research Institute- Site Number : 8400085, Tucson, Arizona
  - Modena Allergy + Asthma- Site Number : 8400021, La Jolla, California
  - Velocity Clinical Research - San Diego- Site Number : 8400024, La Mesa, California
  - Ark Clinical Research- Site Number : 8400097, Long Beach, California
  - Downtown L.A. Research Center- Site Number : 8400080, Los Angeles, California
  - Carbon Health - North Hollywood - NoHo West- Site Number : 8400061, North Hollywood, California
  - Carbon Health - San Mateo - Hillsdale Mall- Site Number : 8400062, San Mateo, California
  - Modena Allergy And Asthma- Site Number : 8400068, Torrance, California
  - Howard University Hospital- Site Number : 8400107, Washington D.C., District of Columbia
  - Helix Biomedics- Site Number : 8400005, Boynton Beach, Florida
  - Beautiful Minds Clinical Research Center- Site Number : 8400019, Cutler Bay, Florida
  - Omega Research Consultants - Debary - North Charles Richard Beall Boulevard- Site Number : 8400082, DeBary, Florida
  - Alfa Medical Research- Site Number : 8400071, Hollywood, Florida
  - Royal Clinical Trials - Inverness- Site Number : 8400067, Inverness, Florida
  - Premier Medical Associates- Site Number : 8400077, Lady Lake, Florida
  - D&H Pompano Research Center- Site Number : 8400072, Margate, Florida
  - Research Institute of South Florida- Site Number : 8400023, Miami, Florida
  - Innovations Biotech- Site Number : 8400044, Miami, Florida
  - Oviedo Medical Research - Site number: 8400091, Oviedo, Florida
  - Tellabio International Research Services- Site Number : 8400083, Pembroke Pines, Florida
  - Avanza Medical Research Center- Site Number : 8400056, Pensacola, Florida
  - Hull and Hull Medical Specialists- Site Number : 8400079, Plantation, Florida
  - Ilumina Medical Research- Site Number : 8400095, Saint Cloud, Florida
  - Private Practice - Dr. David Kavtaradze- Site Number : 8400081, Cordele, Georgia
  - EmVenio Research - Riverdale- Site Number : 8400109, Riverdale, Georgia
  - Christie Clinic in Champaign on University- Site Number : 8400003, Champaign, Illinois
  - University of Kansas Medical Center- Site Number : 8400105, Kansas City, Kansas
  - Velocity Clinical Research - Rockville- Site Number : 8400036, Rockville, Maryland
  - Javara - Privia Medical Group - Silver Spring Lockwood- Site Number : 8400042, Silver Spring, Maryland
  - University of Michigan Health System - Ann Arbor- Site Number : 8400014, Ann Arbor, Michigan
  - Clarkston Medical Group- Site Number : 8400054, Clarkston, Michigan
  - Javara - Mankato Clinic- Site Number : 8400001, Mankato, Minnesota
  - Mayo Clinic in Rochester - Minnesota- Site Number : 8400057, Rochester, Minnesota
  - Hannibal Regional Healthcare System- Site Number : 8400078, Hannibal, Missouri
  - Icahn School of Medicine at Mount Sinai (ISMMS) - Mount Sinai Doctors- Site Number : 8400069, New York, New York
  - Pioneer Clinical Research - New York- Site Number : 8400092, New York, New York
  - Piedmont Healthcare - Family Medicine- Site Number : 8400064, Statesville, North Carolina
  - Cleveland Clinic - Cleveland- Site Number : 8400106, Cleveland, Ohio
  - Asthma & Allergy Center - Toledo- Site Number : 8400020, Toledo, Ohio
  - OK Clinical Research- Site Number : 8400060, Edmond, Oklahoma
  - Clinical Research Associates of Central PA- Site Number : 8400013, DuBois, Pennsylvania
  - Thomas Jefferson University Hospital- Site Number : 8400110, Philadelphia, Pennsylvania
  - ADAC Research- Site Number : 8400070, Greenville, South Carolina
  - Orion Clinical Research, Austin, Texas
  - South Texas Medical Research Institute - TTS Research- Site Number : 8400015, Boerne, Texas
  - Epic Medical Research - De Soto- Site Number : 8400051, DeSoto, Texas
  - Axsendo Clinical Research - Houston- Site Number : 8400065, Houston, Texas
  - Radiance Clinical Research - Lampasas - West Avenue East- Site Number : 8400087, Lampasas, Texas
  - Metroplex Pulmonary and Sleep Center- Site Number : 8400012, McKinney, Texas
  - STAAMP Research - San Antonio- Site Number : 8400059, San Antonio, Texas
  - Bandera Family Health Care - San Antonio- Site Number : 8400049, San Antonio, Texas
  - Javara - San Marcos - Redwood Road- Site Number : 8400040, San Marcos, Texas
  - Javara - Privia Medical Group North Texas - Stephenville- Site Number : 8400038, Stephenville, Texas
  - Simcare Medical Research- Site Number : 8400102, Sugar Land, Texas
  - Children's Wisconsin- Site Number : 8400073, Milwaukee, Wisconsin
- Argentina (16):
  - Investigational Site Number : 0320007, Berazategui, Buenos Aires
  - Investigational Site Number : 0320011, La Plata, Buenos Aires
  - Investigational Site Number : 0320013, Lobos, Buenos Aires
  - Investigational Site Number : 0320006, Rosario, Santa Fe Province
  - Investigational Site Number : 0320010, Rosario, Santa Fe Province
  - Investigational Site Number : 0320016, Rosario, Santa Fe Province
  - Investigational Site Number : 0320003, San Miguel de Tucumán, Tucumán Province
  - Investigational Site Number : 0320005, Buenos Aires
  - Investigational Site Number : 0320012, Buenos Aires
  - Investigational Site Number : 0320002, Buenos Aires
  - Investigational Site Number : 0320001, Buenos Aires
  - Investigational Site Number : 0320004, Buenos Aires
  - Investigational Site Number : 0320008, Corrientes
  - Investigational Site Number : 0320014, Mendoza
  - Investigational Site Number : 0320015, Mendoza
  - Investigational Site Number : 0320009, Santa Fe
- Belgium (3):
  - Investigational Site Number : 0560001, Ghent
  - Investigational Site Number : 0560003, Liège
  - Investigational Site Number : 0560002, Mechelen
- Brazil (6):
  - Associacao Proar- Site Number : 0760002, Salvador, Estado de Bahia
  - Universidade Federal de Goias- Site Number : 0760011, Goiânia, Goiás
  - Hospital de Clinicas da Universidade Federal do Parana- Site Number : 0760006, Curitiba, Paraná
  - Hospital São Lucas da PUCRS - Porto Alegre - Avenida Ipiranga- Site Number : 0760001, Porto Alegre, Rio Grande do Sul
  - WM Pesquisas Clínicas em Doenças Respiratórias- Site Number : 0760003, Porto Alegre, Rio Grande do Sul
  - Incor - Instituto do Coracao- Site Number : 0760004, São Paulo
- Canada (8):
  - Investigational Site Number : 1240011, Kelowna, British Columbia
  - Investigational Site Number : 1240012, West Vancouver, British Columbia
  - Investigational Site Number : 1240013, Ajax, Ontario
  - Investigational Site Number : 1240003, Guelph, Ontario
  - Investigational Site Number : 1240006, Stoney Creek, Ontario
  - Investigational Site Number : 1240008, Toronto, Ontario
  - Investigational Site Number : 1240014, Montreal, Quebec
  - Investigational Site Number : 1240002, Sherbrooke, Quebec
- Chile (10):
  - Investigational Site Number : 1520002, Talca, Maule Region
  - Investigational Site Number : 1520009, Lo Barnechea, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520010, Recoleta, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520006, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520001, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520003, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520005, Quillota, Región de Valparaíso
  - Investigational Site Number : 1520004, Viña del Mar, Región de Valparaíso
  - Investigational Site Number : 1520007, Viña del Mar, Región de Valparaíso
  - Investigational Site Number : 1520008, Concepción, Región del Biobío
- China (40):
  - Investigational Site Number : 1560027, Beijing
  - Investigational Site Number : 1560005, Changchun
  - Investigational Site Number : 1560021, Chengde
  - Investigational Site Number : 1560039, Chengdu
  - Investigational Site Number : 1560028, Foshan
  - Investigational Site Number : 1560010, Guangzhou
  - Investigational Site Number : 1560033, Guangzhou
  - Investigational Site Number : 1560037, Guiyang
  - Investigational Site Number : 1560042, Hangzhou
  - Investigational Site Number : 1560009, Hebei
  - Investigational Site Number : 1560040, Hefei
  - Investigational Site Number : 1560006, Hohhot
  - Investigational Site Number : 1560007, Hohhot
  - Investigational Site Number : 1560029, Huizhou
  - Investigational Site Number : 1560011, Huizhou
  - Investigational Site Number : 1560025, Jiazhuang
  - Investigational Site Number : 1560034, Jinan
  - Investigational Site Number : 1560038, Jinan
  - Investigational Site Number : 1560030, Lanzhou
  - Investigational Site Number : 1560018, Luoyang
  - Investigational Site Number : 1560003, Nanchang
  - Investigational Site Number : 1560014, Ningbo
  - Investigational Site Number : 1560001, Shanghai
  - Investigational Site Number : 1560043, Shanghai
  - Investigational Site Number : 1560016, Shenyang
  - Investigational Site Number : 1560019, Suzhou
  - Investigational Site Number : 1560008, Suzhou
  - Investigational Site Number : 1560017, Taiyuan
  - Investigational Site Number : 1560035, Taiyuan
  - Investigational Site Number : 1560002, Tianjin
  - Investigational Site Number : 1560013, Tianjin
  - Investigational Site Number : 1560022, Wuhan
  - Investigational Site Number : 1560036, Xi'an
  - Investigational Site Number : 1560032, Xi'an
  - Investigational Site Number : 1560044, Xianyang
  - Investigational Site Number : 1560012, Xuzhou
  - Investigational Site Number : 1560047, Yangzhou
  - Investigational Site Number : 1560023, Zhengzhou
  - Investigational Site Number : 1560026, Zhengzhou
  - Investigational Site Number : 1560045, Zigong
- Denmark (2):
  - Investigational Site Number : 2080001, Hvidovre
  - Investigational Site Number : 2080002, Vejle
- France (6):
  - Investigational Site Number : 2500007, Amiens
  - Investigational Site Number : 2500004, Lyon
  - Investigational Site Number : 2500003, Montpellier
  - Investigational Site Number : 2500005, Pessac
  - Investigational Site Number : 2500001, Strasbourg
  - Investigational Site Number : 2500002, Toulouse
- Germany (8):
  - Investigational Site Number : 2760006, Ahrensburg
  - Investigational Site Number : 2760002, Bendorf
  - Investigational Site Number : 2760007, Berlin
  - Investigational Site Number : 6420001, Düsseldorf
  - Investigational Site Number : 2760004, Frankfurt
  - Investigational Site Number : 2760008, Frankfurt
  - Investigational Site Number : 2760001, Leipzig
  - Investigational Site Number : 2760005, Mainz
- Hungary (6):
  - Investigational Site Number : 3480006, Debrecen
  - Investigational Site Number : 3480002, Gödöllő
  - Investigational Site Number : 3480003, Hajdúnánás
  - Investigational Site Number : 3480004, Mosonmagyaróvár
  - Investigational Site Number : 3480005, Pécs
  - Investigational Site Number : 3480001, Püspökladány
- Investigational Site Number : 2500006, Mumbai, India
- Israel (6):
  - Investigational Site Number : 3760006, Haifa
  - Investigational Site Number : 3760003, Jerusalem
  - Investigational Site Number : 3760002, Jerusalem
  - Investigational Site Number : 3760005, Petah Tikva
  - Investigational Site Number : 3760001, Rehovot
  - Investigational Site Number : 3760004, Tel Aviv
- Italy (12):
  - Investigational Site Number : 3800008, Torette, Ancona
  - Investigational Site Number : 3800006, Monserrato, Cagliari
  - Investigational Site Number : 3800001, Cona, Ferrara
  - Investigational Site Number : 3800009, Genoa, Genova
  - Investigational Site Number : 3800004, Milan, Milano
  - Investigational Site Number : 3800003, Rozzano, Milano
  - Investigational Site Number : 3800010, Rome, Roma
  - Investigational Site Number : 3800012, Tradate, Varese
  - Investigational Site Number : 3800007, Bergamo
  - Investigational Site Number : 3800005, Modena
  - Investigational Site Number : 3800013, Palermo
  - Investigational Site Number : 3800011, Reggio Emilia
- Japan (3):
  - Investigational Site Number : 3920002, Shinagawa, Tokyo
  - Investigational Site Number : 3920001, Ube, Yamaguchi
  - Investigational Site Number : 3920004, Tokyo
- Mexico (5):
  - Investigational Site Number : 4840001, Guadalajara, Jalisco
  - Investigational Site Number : 4840007, Guadalajara, Jalisco
  - Investigational Site Number : 4840005, Monterrey, Nuevo León
  - Investigational Site Number : 4840006, San Juan del Río, Querétaro
  - Investigational Site Number : 4840002, Chihuahua City
- Poland (7):
  - Investigational Site Number : 6160005, Poznan, Greater Poland Voivodeship
  - Investigational Site Number : 6160001, Poznan, Greater Poland Voivodeship
  - Investigational Site Number : 6160008, Lodz, Lódzkie
  - Investigational Site Number : 6160002, Bialystok, Podlaskie Voivodeship
  - Investigational Site Number : 6160004, Chęciny
  - Investigational Site Number : 6160009, Katowice
  - Investigational Site Number : 6160003, Ostrowiec Świętokrzyski, Świętokrzyskie Voivodeship
- Investigational Site Number : 6420002, Cluj-Napoca, Romania
- South Africa (6):
  - Investigational Site Number : 7100004, Benoni
  - Investigational Site Number : 7100005, Benoni
  - Investigational Site Number : 7100002, Cape Town
  - Investigational Site Number : 7100003, Durban
  - Investigational Site Number : 7100006, Durban
  - Investigational Site Number : 7100007, Johannesburg
- Spain (16):
  - Investigational Site Number : 7240005, Santiago de Compostela, A Coruña [La Coruña]
  - Investigational Site Number : 7240010, Badalona, Barcelona [Barcelona]
  - Investigational Site Number : 7240009, Barcelona, Barcelona [Barcelona]
  - Investigational Site Number : 7240015, Barcelona, Barcelona [Barcelona]
  - Investigational Site Number : 7240017, Santander, Cantabria
  - Investigational Site Number : 7240016, Girona, Girona [Gerona]
  - Investigational Site Number : 7240018, Benalmádena, Málaga
  - Investigational Site Number : 7240013, Madrid
  - Investigational Site Number : 7240008, Madrid
  - Investigational Site Number : 7240011, Madrid
  - Investigational Site Number : 7240002, Madrid
  - Investigational Site Number : 7240007, Madrid
  - Investigational Site Number : 7240004, Málaga
  - Investigational Site Number : 7240006, Málaga
  - Investigational Site Number : 7240001, Palma
  - Investigational Site Number : 7240014, Seville
- Sweden (3):
  - Investigational Site Number : 7520003, Gothenburg
  - Investigational Site Number : 7520002, Lund
  - Investigational Site Number : 7520001, Solna
- Taiwan (7):
  - Investigational Site Number : 1580002, Hualien City
  - Investigational Site Number : 1580005, Kaohsiung City
  - Investigational Site Number : 1580006, Taichung
  - Investigational Site Number : 1580007, Taichung
  - Investigational Site Number : 1580004, Taipei
  - Investigational Site Number : 1580003, Taipei
  - Investigational Site Number : 1580001, Taoyuan
- Turkey (Türkiye) (3):
  - Investigational Site Number : 7920003, Kayseri
  - Investigational Site Number : 7920002, Kırıkkale
  - Investigational Site Number : 7920001, Mersin
- United Kingdom (7):
  - Investigational Site Number : 8260007, Corby, Northamptonshire
  - Investigational Site Number : 8260006, Nottingham, Nottinghamshire
  - Investigational Site Number : 8260008, Oxford, Oxfordshire
  - Investigational Site Number : 8260005, Barnsley
  - Investigational Site Number : 8260003, Bradford
  - Investigational Site Number : 8260009, Hillingdon
  - Investigational Site Number : 8260001, London

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: ACT18301 Plain Language Results Summary — https://sanofi.trialsummaries.com/Study/StudyDetails?id=26271&tenant=MT_SNY_9011